CLINICAL TRIAL: NCT02625896
Title: Free Fall Acrobatics to Reduce Neck Loads During Parachute Opening Shock: Evaluation of an Intervention.
Acronym: ACROPOSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Anton Westman, MD PhD, Karolinska Institutet
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: CIF FO2015-0005.; CIF D2014-0021 (Other: The Swedish National Centre for Research in Sports (CIF))
Record Dates: First submitted 2015-12-07; First posted 2015-12-09 (Estimated); Last update posted 2018-10-30 (Actual); Status verified 2018-10

CONDITIONS: Pain; Athletic Injuries; Whiplash Injuries; Biomechanical Lesion, Unspecified
Keywords: Aviation; Parachuting
MeSH Terms: conditions — Pain; Athletic Injuries; Whiplash Injuries | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): A sequence of free fall manoeuvres performed using the human body: A free fall velocity reduction prior to main parachute deployment followed by a head high body attitude prior to main parachute extraction.
  Interventions: Behavioral: Intervention
- Control (No Intervention): Normal main parachute extraction performed in a manner that is typical for the study participant.

INTERVENTIONS:
Behavioral: Intervention — Standard skydive from 4 000 m above mean sea level (AMSL) following standard safety recommendations and procedures including, if necessary, standard reserve parachute activation procedures. If necessary for safety, participants are asked to immediately leave the study at will. At 1 500 m AMSL, the participant is asked to begin to slow down the fall rate by increasing the body surface area to the relative wind. At no lower than 1 200 m AMSL, the participant is asked to deploy the main parachute. At main parachute deployment, while maintaining a stable body position with shoulders level to the horizon and unaltered heading, the participant is asked to increase the pitch angle of the long body axis attitude, raising the head, shoulders, and upper body up from the flat belly-to-relative-wind plane to a head-high body position, using any free fall technique the participant is comfortable with - as long as there is NO RISK for an unintentional backflip.
  Arms: Intervention

SUMMARY:
This study aims to evaluate the use of an aerial human body manoeuvre to reduce the biomechanical load on the neck of a parachutist during the parachute opening, in order to create a basis for future prevention of skydiver neck pain in the parachutist population.

DETAILED DESCRIPTION:
Elevated neck pain prevalence among skydivers is associated with exposure to repeated parachute openings. The parachute opening shock (POS) is a sudden and brutal deceleration of a human being. In skydiving (sport parachuting from aircraft), it slows a free falling skydiver from a velocity >200 km/h to <30 km/h within a few seconds. POS deceleration magnitudes 9-12 times Earth's gravitational acceleration (a dimensionless ratio denoted G) have been measured. These hard openings were painful, and a number of very hard openings have generated injuries visible to health care systems. During subjectively normal openings, decelerations measured on the human neck exceed 4 G with initial onset rates (jerks) exceeding 20 G/s. Considering that active skydivers may do ten jumps per day and may accumulate well over a thousand jumps during a parachuting career, these are problematic values. Fighter pilots have suffered neck pain after less accelerative exposure. In the Swedish skydiving population, the neck pain prevalence is 45%, to be compared with a general population estimate of 37%. Recently published data show that skydiver neck muscles are under excessive strain during POS, and data from our group suggest POS as composed of biomechanically discrete phases. A first phase contains an initial jerk in ventral to dorsal direction, i.e. "pulled backwards", denoted negative Gx, when the skydiver is rapidly rotated from a prone belly-to-earth body position to an upright position. During this phase, the moment arm from the center of mass of the head to the parachute connection point at the shoulders is long and likely to yield a high torque in the neck. The second phase, denoted positive Gz, contains the bulk of POS-deceleration directed caudally to cranially. Entering the second phase with the neck flexed forward from the jerk would put the neck muscles in a clear disadvantage.

In a sport, it would seem desirable to prevent injuries by the way the sport is practiced. A number of techniques to reduce POS neck loads have been suggested among athletes, two of which are biomechanically appealing: Reducing parachute deployment airspeed and positioning the human body head high prior to main parachute extraction. Whether these techniques actually reduce neck loads during POS has not been systematically evaluated. From an empirically determined relation between maximum POS deceleration and free fall velocity, it can be calculated that a decrease in velocity from 220 km/h to 190 km/h may reduce the maximum deceleration and thereby (constant mass) force 25%. Such a velocity reduction is possible using the human body only. Our static anthropometrical assessments suggest that, unless a flexion forward of the head occurs, pitching up the body head high to an angle of 45 degrees from the flat-belly-to-relative-wind plane may reduce the head-neck lever arm 30%. Thus, a successful combination of velocity reduction and head-neck lever arm reduction holds the promise of an approximately halved torque in the neck during POS. Such a substantial mechanical change can be hypothesized to have biological effects.

The intervention protocol is based on observational data and static anthropometrical calculations and inspired by anecdotal information. It has been systematically validated by subject matter experts, and the results of this validation has been published. The intervention is conceived as a combination of velocity reduction and head-neck lever arm reduction, main outcome variables being magnitudes of decelerations and jerks, expressed in G and G/s, respectively, and research subjects being experienced skydivers completing two consecutive skydives on the same day with random ordering (one being the control jump and one being the intervention jump).

Based on an estimated real-world 30% effect size and a desired 0.9 power level, sample size calculation suggest 16 subjects as sufficient for parametric analyses. To allow for dropout, the sample size will be increased to 20 subjects. Thus, twenty highly experienced skydivers will be recruited to the study, to perform the two consecutive terminal velocity skydives on the same day. Their demographics and background data will be obtained with use of a validated web-based questionnaire for skydivers. The test subjects will be recruited through electronic fora, including e-mail lists, for highly experienced skydivers. They will use their own sport parachute systems packed and maintained by themselves. The rationale for this is to maintain typical and comfortable conditions for each subject, whereas an unfamiliar system may introduce undesired psychomotor confounders, and also to maintain a high degree of external validity (as compared to using only one type of standardized parachute).

A detailed description of the planned measuring instrumentation has been published separately. The equipment setup in its entirety is approved for aerial use by the National Safety Officer of the Swedish Parachute Association. Multiple triaxial accelerometers are used to measure decelerations and jerks, and videography to record complex movements, including the parachute opening and head motion. Altitude and falling speed data will be collected with barometric and Global Positioning System (GPS) altimetry, using state-of-the-art skydiving devices.

Two consecutive skydives from 4000 m altitude will be completed by each subject on the same day; one being the control jump and one being the intervention jump. For safety reasons, main parachute terminal velocity deployment altitude will be elevated above normal and high-speed landings forbidden. In one of the two skydives, the test subject will perform an intervention consisting of a sequence of free fall manoeuvres performed using the human body: A free fall velocity reduction prior to main parachute deployment followed by a head high body attitude prior to main parachute extraction. Details of the manoeuvres will be given to the test subject in a written instruction.

This study will use a cross-over, within-subject, repeated measures design with random ordering of performing intervention jump or "ordinary" jump in the first jump of two. Computerized randomization will be performed in blocks, i.e. to have equal numbers of subjects starting with intervention jump vs. control jump in a block of every four subjects. A detailed description of the planned methodology for treatment and analysis of data has been published separately. Repeated within group measures ANOVA is planned to be used to measure effects, and regression used to test for relationships.

The results of this study are expected to contribute to a basis for future prevention of neck pain among skydivers, which is known to have a relation to repeated parachute opening exposure. In work addressing this health problem, our study may create a logical fork with important future implications. From static biomechanics and theoretical calculations, the planned intervention holds the promise of a halved torque in the neck during parachute opening. Though real-world results may not show such an impressive effect, it is important to examine this assumption; if it can be demonstrated to have some merit, further large-scale population studies and implementation would seem warranted, possibly offering an elegant solution to a widespread health problem in this population. If, on the other hand, the planned intervention can be demonstrated to have little or no effect on its biomechanical outcome variables, doubt will be cast upon the conventional wisdom skydiver good advice upon which it is based, shifting future attention more pointedly towards manufacturers of parachute systems.

This study will be conducted in Swedish airspace in cooperation with and under the supervision of the National Safety Officer of the Swedish Parachute Association. All safety resources for sport parachuting available within the Swedish Parachute Association will be employed. This study will be conducted in compliance with the Declaration of Helsinki. All subjects will receive oral and written information about the study, including safety aspects (e.g., agreeing not to perform high-speed landings during the study), and sign a written consent to participate. All subjects will be informed that they can end the study participation at any time.

ELIGIBILITY:
Inclusion Criteria:

* Holders of the highest parachute certification (level D) in the Swedish Parachute Association

Exclusion Criteria:

* Ongoing neck problems
* Pregnancy
* Unwillingness to follow the safety regulations of the study
* Known patch allergy
* Participation in another concurrent biomedical study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2017-06-17 (Actual); Primary Completion 2018-10-14 (Actual); Study Completion 2018-10-14 (Actual)

PRIMARY OUTCOMES:
Magnitudes of decelerations | 10 seconds
  Multidirectional accelerations during ram-air parachute openings expressed in terms of multiples of Earth's gravitational acceleration g using the dimensionless ratio G.
Magnitudes of jerks | 10 seconds
  Multidirectional rates of changes of accelerations during ram-air parachute openings expressed in G per second.

CONTACTS AND LOCATIONS:
Overall Officials: Anton Westman, MD PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Stockholm, Sweden

REFERENCES:
- [Background] Westman A, Bjornstig U. Injuries in Swedish skydiving. Br J Sports Med. 2007 Jun;41(6):356-64; discussion 364. doi: 10.1136/bjsm.2006.031682. Epub 2007 Jan 15. PMID 17224436
- [Background] Westman A, Sjoling M, Lindberg A, Bjornstig U. The SKYNET data: demography and injury reporting in Swedish skydiving. Accid Anal Prev. 2010 Mar;42(2):778-83. doi: 10.1016/j.aap.2009.11.013. Epub 2009 Dec 31. PMID 20159107
- [Background] Nilsson J, Friden C, Buren V, Westman A, Lindholm P, Ang BO. Musculoskeletal pain and related risks in skydivers: a population-based survey. Aviat Space Environ Med. 2013 Oct;84(10):1034-40. doi: 10.3357/asem.3570.2013. PMID 24261055
- [Background] Gladh K, Ang BO, Lindholm P, Nilsson J, Westman A. Decelerations and muscle responses during parachute opening shock. Aviat Space Environ Med. 2013 Nov;84(11):1205-10. doi: 10.3357/asem.3637.2013. PMID 24279237
- [Background] Lo Martire R, Gladh K, Westman A, Lindholm P, Nilsson J, Ang BO. Neck muscle activity in skydivers during parachute opening shock. Scand J Med Sci Sports. 2016 Mar;26(3):307-16. doi: 10.1111/sms.12428. Epub 2015 Mar 10. PMID 25754941
- [Derived] Westman A, Ang BO. Free Fall Acrobatics to Reduce Neck Loads During Parachute Opening Shock: Evaluation of an Intervention (ACROPOSE). BMJ Open Sport Exerc Med. 2016 Apr 26;2(1):e000108. doi: 10.1136/bmjsem-2015-000108. eCollection 2016. PMID 27900175